CLINICAL TRIAL: NCT04586400
Title: Genotype-Phenotype Correlation in Patients With Chromosome 9 P Minus Syndrome
Brief Title: Chromosome 9 P Minus Syndrome
Status: Recruiting | Type: Observational
Sponsor: Washington University School of Medicine (Other)
Collaborators: Dickson, Patricia I., M.D. (Individual); Milbrandt, Jeffrey, MD, PhD (Unknown); Mitra, Rob, PhD (Unknown); Turner, Tychele, PhD (Unknown)
Responsible Party: Sponsor
Other Study IDs: 201706062
Record Dates: First submitted 2020-10-06; First posted 2020-10-14 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Chromosome 9P Deletion Syndrome; 9p Minus Syndrome; Alfi Syndrome; 9P Monosomy; 9P Partial Monosomy Syndrome
MeSH Terms: conditions — Chromosome 9p Deletion Syndrome; Chromosome 9, partial monosomy 9p

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva, blood or skin biopsy samples may be obtained in this study. A study team member will discuss this with you.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Patients with deletion of chromosome 9 P are rare (~200 in the medical literature) and have a diverse set of phenotypic characteristics. We propose using state of the art genome sequencing methods to define the location and size of the deleted portion of chromosome 9 P as well as the genetic background in affected patients (whole genome sequencing) and correlate the genes in the deleted portion of chromosome 9 P with specific phenotypic characteristics of each patient. Enrolled participants will be asked to complete a detailed questionnaire, complete a medical release form, and provide a biospecimen sample.

ELIGIBILITY:
Inclusion Criteria:

* Having 9P minus syndrome/ deletions on the 9th chromosome
* Parents and siblings of affected individuals may also be included to determine contribution of genetic background to phenotypic characteristics

Exclusion Criteria:

* No exclusion criteria for either affected individuals or their parents or siblings.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The Principal Investigator and members of the study team in collaboration with the 9 P Minus Network (http://9pminus.org/), Unique (https://www.rarechromo.org/), and other members of the 9 P Minus community will identify candidate participants with 9 P minus syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2017-06-27 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Genotypic and Phenotypic Correlation | As enrollment increases the team hopes to have preliminary results by 2022
  By use of demographic and genetic material we hope to gain a better understanding between the deletion on the short arm of the 9th chromosome and the features presented.

CONTACTS AND LOCATIONS:
Overall Officials: F. S Cole, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No
The study was created to have a better understanding of 9P minus syndrome. The team will educate participants regarding their genetic testing but this is not intended to influence medical decisions.